CLINICAL TRIAL: NCT06956677
Title: Usability and Effectiveness of a Novel Bilateral Upper Limb Training Device for Stroke Patients With Hemiparesis: A Preliminary Study
Acronym: Synslai
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202301097A3
Record Dates: First submitted 2025-04-24; First posted 2025-05-04 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2023-09

CONDITIONS: The Effectiveness of Novel Rehabilitation Device on Upper Limb Impairment Among Patients With Stroke
Keywords: Stroke; Hemiparesis; Usability; Bilateral Training; Upper Extremity Rehabilitation
MeSH Terms: conditions — Stroke; Paresis

STUDY DESIGN:
Intervention Model Description: An investigator analyzed inclusion and exclusion criteria and assigned participants to one of the groups. Participants were randomly allocated to either the experimental group or the control group. Randomization and group allocation was performed by a research assistant using a computer-generated randomization sequence to ensure unbiased allocation. Each intervention was conducted over a 3-week period, consisting of 10 to 15 sessions.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): Intervention includes 30 minutes of UE functional training and 1 hour of conventional occupational therapy.
  Interventions: Other: The UE functional training; Other: Conventional occupational therapy
- Experimental group (Experimental): Intervention consists of 30 minutes of novel UE rehabilitation device training and 1 hour of conventional occupational therapy.
  Interventions: Device: Novel UE rehabilitation device training; Other: Conventional occupational therapy

INTERVENTIONS:
Device: Novel UE rehabilitation device training — The novel UE rehabilitation device training includes the single-joint exercise and dual-joint exercise, each performed 20 repetitions per set, for a total of 5 sets with 30-second rest intervals between sets.
  Arms: Experimental group
Other: The UE functional training — The UE functional training focuses on the affected arm, incorporating exercises such as push-pull boxes (standing or seated), alternating push-pull boxes, and hand-crank exercises.
  Arms: Control group
Other: Conventional occupational therapy — Conventional occupational therapy

SUMMARY:
Background and Study Aims Stroke is a leading cause of long-term disability worldwide, affecting millions of individuals each year. After experiencing a stroke, many patients face challenges with their upper limbs, resulting in difficulties in performing daily activities. This study aims to evaluate a new rehabilitation device designed to assist stroke patients with hemiparesis (weakness on one side of the body) in improving their upper limb function. The goal is to determine if this device can effectively support recovery while providing an affordable and accessible option for rehabilitation.

Who Can Participate? This study is open to adults aged between 18 and 70 years, regardless of sex. To participate, individuals must have a confirmed diagnosis of hemiplegic stroke, which means they must experience weakness in one side of the body. Participants should have had their stroke within the last 12 months and must be able to follow simple commands. Those with cognitive impairments, other neurological disorders, certain orthopedic conditions affecting the upper limb, or active skin issues will not be eligible.

What Does the Study Involve? Participants in this study will be randomly assigned to two groups: one group will use the new rehabilitation device, while the other will receive conventional occupational therapy. Both groups will undergo an assessment before and after the intervention to measure their improvement in upper limb function. The device encourages exercises that are essential for fostering movement recovery, while the conventional therapy focuses on traditional rehabilitation methods. Participants will have their upper limb function evaluated through established assessment tools to gauge progress.

What Are the Possible Benefits and Risks of Participating? By participating in this study, individuals may experience improvements in their upper limb function, leading to increased independence and enhanced quality of life. Additionally, participants will contribute to valuable research that could improve rehabilitation strategies for future stroke patients. While the rehabilitation device is designed to be safe, some individuals may experience mild discomfort or fatigue from the exercises. However, serious side effects are rare. Participants are encouraged to discuss any concerns with the research team.

Where Is the Study Run From? The study is being conducted at New Taipei Municipal TuCheng Hospital in Taiwan, specifically in the rehabilitation ward, where trained medical professionals oversee the research process.

When Is the Study Starting and How Long Is It Expected to Run For? The study commenced in September 2023 and is expected to continue through November 2024. This timeline allows for recruiting participants and thorough data collection to assess the device's effectiveness.

Who Is Funding the Study? This study does not have external funding and is being conducted independently by the researchers involved. All costs associated with the study, including participant care and device usage, are covered by the resources of the conducting institution.

Who Is the Main Contact?

For more information about this study, please contact:

Kuo-Cheng, Liu Position: Research Coordinator Email address: monhh159@gmail.com

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed stroke diagnosis by imaging, with onset within the past 12 months
2. Age between 18 and 70 years
3. Stable physiological and neurological status (no neurological deterioration and stable vital signs for ≥72 hours; complications resolved or medically managed)
4. Adequate cognitive function to follow at least two-step commands
5. Willingness to provide written informed consent
6. Unilateral upper extremity (UE) hemiplegia
7. Brunnstrom stage > I for proximal UE motor function
8. UE muscle tone < 3 on the Modified Ashworth Scale

Exclusion Criteria:

1. Cognitive impairment
2. Other neurological disorders
3. Orthopedic conditions affecting the UE
4. Active or non-healed dermatological lesions

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2023-09-05 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Fugl-Meyer Assessment for Upper Extremity | Outcome measurements were performed at three stages: before and after (immediately following the final session) the intervention.
  This assessment captures motor recovery across four specific domains: Part A (proximal upper limb-shoulder, elbow, and forearm), Part B (wrist), Part C (hand), and Part D (coordination and speed). The full scale ranges from 0 to 66 and the higher scores represent the better outcome.

SECONDARY OUTCOMES:
Brunnstrom stage | Outcome measurements were performed at three stages: before and after (immediately following the final session) the intervention.
  The Brunnstrom scale classifies motor recovery post-stroke into six stages, ranging from flaccid paralysis (Stage I) to near-normal voluntary control (Stage VI), and the higher stage represent the better outcome.
Modified Ashworth scale | Outcome measurements were performed at three stages: before, during (after the 5th training session), and after (immediately following the final session) the intervention.
  This scale assesses the severity of muscle spasticity by quantifying resistance to passive movement on a scale from 0 (no increase in tone) to 4 (rigid in flexion or extension) and the higer scores represent the worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- New Taipei Municipal TuCheng Hospital, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
The datasets generated during and/or analysed during the current study were available upon request from
  * Contact Name and Email Address: Dr. Kuo-Cheng Liu, email: monhh159@gmail.com
  * Type of Data Shared: Individual participant data (IPD) including demographic, assessments, interventions.
  * Availability: The dataset will be available upon request after the publication of study results.
  * Access Criteria: Researchers can request data by providing a brief description of their intended analysis, which should align with stroke rehabilitation research objectives.
  * Consent from Participants: Informed consent was obtained.
  * Anonymization Comments: Data will be anonymized to protect participant identities.
  * Ethical or Legal Restrictions: Following ethical guidelines and IRB requirements will guide the data-sharing process.
  * Other Comments: Participants' consents specify academic and appropriate use of data.
Supporting Information: Study Protocol

REFERENCES:
- [Result] Sahu RK, Gugnani A, Ahluwalia R. Short-term effectiveness of trunk and bimanual hand training on upper limb motor recovery and function in stroke patients. International journal of health sciences. 05/15 2022;6(S1):10058-10071. doi:10.53730/ijhs.v6nS1.7384
- [Result] Julien M, Laffont I, Bonnin H-Y, Liesjet V, Mottet D. Bimanual Coordination Being Efficient Around Two Months After Stroke: A Key Recovery Moment for Starting Bimanual Rehabilitation Protocols? BIO Web of Conferences. 12/01 2011;1doi:10.1051/bioconf/20110100062
- [Result] Metrot J, Mottet D, Hauret I, van Dokkum L, Bonnin-Koang HY, Torre K, Laffont I. Changes in bimanual coordination during the first 6 weeks after moderate hemiparetic stroke. Neurorehabil Neural Repair. 2013 Mar-Apr;27(3):251-9. doi: 10.1177/1545968312461072. Epub 2012 Nov 7. PMID 23135767
- [Result] Ma D, Li X, Xu Q, Yang F, Feng Y, Wang W, Huang JJ, Pei YC, Pan Y. Robot-Assisted Bimanual Training Improves Hand Function in Patients With Subacute Stroke: A Randomized Controlled Pilot Study. Front Neurol. 2022 Jul 6;13:884261. doi: 10.3389/fneur.2022.884261. eCollection 2022. PMID 35873779
- [Result] Shahid J, Kashif A, Shahid MK. A Comprehensive Review of Physical Therapy Interventions for Stroke Rehabilitation: Impairment-Based Approaches and Functional Goals. Brain Sci. 2023 Apr 25;13(5):717. doi: 10.3390/brainsci13050717. PMID 37239189
- [Result] Nair KPST, A B. Stroke rehabilitation : traditional and modern approaches. 2002;
- [Result] Tan CO. Is remote rehabilitation after stroke as effective as conventional therapy? Neurology. 2020 Oct 27;95(17):e2462-e2464. doi: 10.1212/WNL.0000000000010839. No abstract available. PMID 33106363
- [Result] Langhorne P, Legg L. Evidence behind stroke rehabilitation. J Neurol Neurosurg Psychiatry. 2003 Dec;74 Suppl 4(Suppl 4):iv18-iv21. doi: 10.1136/jnnp.74.suppl_4.iv18. No abstract available. PMID 14645462
- [Result] Johnson MJ, Rai R, Barathi S, Mendonca R, Bustamante-Valles K. Affordable stroke therapy in high-, low- and middle-income countries: From Theradrive to Rehab CARES, a compact robot gym. J Rehabil Assist Technol Eng. 2017 Jun 1;4:2055668317708732. doi: 10.1177/2055668317708732. eCollection 2017 Jan-Dec. PMID 31186929
- [Result] Mehrholz J, Pohl M, Platz T, Kugler J, Elsner B. Electromechanical and robot-assisted arm training for improving activities of daily living, arm function, and arm muscle strength after stroke. Cochrane Database Syst Rev. 2018 Sep 3;9(9):CD006876. doi: 10.1002/14651858.CD006876.pub5. PMID 30175845
- [Result] Poli P, Morone G, Rosati G, Masiero S. Robotic technologies and rehabilitation: new tools for stroke patients' therapy. Biomed Res Int. 2013;2013:153872. doi: 10.1155/2013/153872. Epub 2013 Nov 20. PMID 24350244
- [Result] Trombly CA, Ma HI. A synthesis of the effects of occupational therapy for persons with stroke, Part I: Restoration of roles, tasks, and activities. Am J Occup Ther. 2002 May-Jun;56(3):250-9. doi: 10.5014/ajot.56.3.250. PMID 12058514
- [Result] Paci M, Nannetti L, Casavola D, Lombardi B. Differences in motor recovery between upper and lower limbs: does stroke subtype make the difference? Int J Rehabil Res. 2016 Jun;39(2):185-7. doi: 10.1097/MRR.0000000000000172. PMID 27096715
- [Result] Parker VM, Wade DT, Langton Hewer R. Loss of arm function after stroke: measurement, frequency, and recovery. Int Rehabil Med. 1986;8(2):69-73. doi: 10.3109/03790798609166178. PMID 3804600
- [Result] McCrea PH, Eng JJ, Hodgson AJ. Biomechanics of reaching: clinical implications for individuals with acquired brain injury. Disabil Rehabil. 2002 Jul 10;24(10):534-41. doi: 10.1080/09638280110115393. PMID 12171643
- [Result] Feigin VL, Brainin M, Norrving B, Martins S, Sacco RL, Hacke W, Fisher M, Pandian J, Lindsay P. World Stroke Organization (WSO): Global Stroke Fact Sheet 2022. Int J Stroke. 2022 Jan;17(1):18-29. doi: 10.1177/17474930211065917. PMID 34986727

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-07-03): https://cdn.clinicaltrials.gov/large-docs/77/NCT06956677/Prot_SAP_000.pdf